CLINICAL TRIAL: NCT04818190
Title: DIEP Flap Sensory Recovery Following Direct Neurotization in Breast Reconstruction - A Blinded Prospective Study
Brief Title: DIEP (Deep Inferior Epigastric Artery Perforator) Flap Sensory Recovery Following Neurotization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HS24687
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-03

CONDITIONS: Sensitisation
Keywords: breast reconstruction; sensory recovery; DIEP reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIEP reconstruction, no neurotization (No Intervention): DIEP reconstruction No sensory neurotization
- DIEP reconstruction, neurotization (Experimental): DIEP reconstruction With sensory neurotization
  Interventions: Procedure: Sensory neurotization

INTERVENTIONS:
Procedure: Sensory neurotization — The donor nerve is a cutaneous nerve that is identified with the most inferior lateral perforator vessels. The nerve is then dissected for neurotization and divided at the level of the fascia where it is a pure sensory nerve. The recipient intercostal nerve is usually easily identified in the third intercostal space during the dissection of the internal mammary artery and vein. The anterior branch of the third intercostal nerve can usually be found at the junction of the inferior portion of the third rib and the sternum, approximately 80% of the time. The nerve is dissected and transected medially. It is then mobilized to give it the longest length possible in preparation for neurotization. Neurotization is performed by coapting the donor nerve to the third anterior intercostal nerve directly with a 9-0 nylon suture in standard fashion.
  Arms: DIEP reconstruction, neurotization

SUMMARY:
The purpose of this study is to compare the sensory return of DIEP flaps with nerve connection to DIEP flaps with no nerve connection to see which is better.

This research is being done because the presence of sensation in a reconstructed breast has been shown to improve patient-related quality of life following mastectomy reconstruction and is an important safety factor for prevention of burns and other flap injuries. Unfortunately, women who have breast skin excised during mastectomy are reconstructed with a traditional DIEP flap that does not restore sensation to the skin.

DETAILED DESCRIPTION:
The Deep Inferior Epigastric Perforator (DIEP) flap is the current standard of care in breast reconstruction. The DIEP flap does not normally have sensation restored. The presence of sensation in a reconstructed breast has been shown to improve patient-rated quality of life following mastectomy and reconstruction and is an important safety factor for prevention of burns and other flap injuries. Unfortunately, women who have breast skin excised during mastectomy are reconstructed with a traditional DIEP flap that does not restore sensation to the skin. As such, the investigators aim to perform a prospective randomized single-blinded trial to evaluate sensory return to DIEP flaps following nerve coaptation.

A blinded, prospective study will be performed involving Manitoban women over 18 years undergoing bilateral breast reconstruction with DIEP flaps. The women will have one breast reconstructed in the standard of care (DIEP flap with no nerve coaptation) and one breast reconstructed with both DIEP flap and sensory nerve coaptation; the side of coaptation will be randomized. Objective sensibility to the breast will be tested pre- and post-operatively (3, 6, 12 months) using the Pressure Specified Sensory Device (PSSD). Patients will also complete the Breast Q questionnaire postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* female subjects older than 18
* scheduled for immediate bilateral breast reconstruction following bilateral non-nipple sparing mastectomy
* using DIEP free flap reconstruction
* with a large skin paddle

Exclusion Criteria:

* pre-operative radiation or chemotherapy was performed
* post-operative radiation or chemotherapy is planned
* reconstruction is performed in a delayed fashion
* a nerve conduit is necessary for nerve coaptation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Sensory recovery to neurotized DIEP flap | 3 months post-operatively
  Sensory recovery measured using Pressure Specified Sensory Device
Sensory recovery to neurotized DIEP flap | 6 months post-operatively
  Sensory recovery measured using Pressure Specified Sensory Device
Sensory recovery to neurotized DIEP flap | 12 months post-operatively
  Sensory recovery measured using Pressure Specified Sensory Device

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Miller, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Science Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04818190/Prot_000.pdf